CLINICAL TRIAL: NCT00935779
Title: Ultra Structure of Peritoneum at Electronic Microscopy in Control Subjects and Patients With Gastric Cancer
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Patricio Burdiles, Hospital Clinico, Universidad de Chile
Other Study IDs: OAIC 043/02
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Stomach Neoplasm
Keywords: Stomach Neoplasms; Peritoneum
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gastric cancer: patients with operable local gastric adenocarcinoma were studied
- Control group: patients operated on for benign diseases served as controls, randomly selected among patients with chronic gastro-esophageal reflux disease who were considered good candidates for antireflux surgery and properly matched in sex and age to study group

SUMMARY:
Peritoneal metastases appear in a great proportion of patients affected by gastric carcinoma. Involved mechanisms are poorly understood though experimentally it has been demonstrated that neoplastic cells exfoliated from primary tumor can only implant and proliferate in areas of damaged peritoneum. Objectives: to study ultra-structure of peritoneal surface by electronic microscopy in control subjects and in patients with early or locally advanced gastric cancer looking for spontaneous changes in peritoneal surface not related with surgical injury.

DETAILED DESCRIPTION:
18 out of 32 cases were eligible for analysis. Four patients operated on for benign diseases served as control and 14 patients with operable local gastric adenocarcinoma (4 mucosa/submucosa/muscular y 10 serosa lesions) were studied. At the beginning of surgery, a 2 x 2 cm. sample from macroscopically normal visceral peritoneum at mesenterium root was carefully obtained, washed with saline and fixed in glutaraldehyde solution. Besides a sample of peritoneal washing fluid was studied to exclude patients with free cancer cells. Peritoneal tissue was fixed during 24 hours and then all samples were evaluated by electronic microscope.

ELIGIBILITY:
Inclusion Criteria:

* patients with operable local gastric adenocarcinoma

Exclusion Criteria:

* previous abdominal surgery
* previous open or blunt abdominal trauma
* history of inflammatory bowel disease or Typhoid Fever, Gallstone disease, chemotherapy or radiotherapy, or any other abdominal condition that could alter peritoneal integrity.
* All other gastric malignancies such as lymphomas, GIST, carcinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with operable local gastric adenocarcinoma consulting to Hospital Clinico, University of Chile during study period.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2002-10; Primary Completion 2004-07 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Burdiles, MD, Principal Investigator — Department of Surgery, Clinical Hospital, University of Chile
Locations (1):
- Department of Surgery, Clinical Hospital, University of Chile, Santiago, Santiago Metropolitan, Chile